CLINICAL TRIAL: NCT05187702
Title: The Effect of Functional Exercise Training on Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Exercise in Hypertension
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-08

CONDITIONS: Hypertension and Balance
Keywords: hypertension; balance; aerobic; otago
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional exercise group and aerobic group (Experimental): Along with functional exercises, aerobic exercises (walking) 3 per week were given.
  Interventions: Other: Functional exersize
- Aerobic Exersize Group (Active Comparator): aerobic exercises (walking) 3 per week were given.
  Interventions: Other: Functional exersize; Other: Aerobic exersize
- Control Group (No Intervention): They continued their daily routine

INTERVENTIONS:
Other: Functional exersize — Participants will be given balance and strengthening exercises covering the balance exercise protocol.
  Arms: Aerobic Exersize Group; Functional exercise group and aerobic group
Other: Aerobic exersize — 60% of the maximum heart rate is given 3 walking eccentricity per week
  Arms: Aerobic Exersize Group

SUMMARY:
It is the ability to keep and maintain the body training balance control center. Dynamic balance is the ability to maintain an individual's static position while the movement and posture are active while static. With aging, it is thought that the system will be applied in practice. Control of cerebral blood flow and synapse, which decreases with advanced age and hypertension, continues. In addition to slowing down in mental functions such as memory and learning, it progresses and accelerates in the sense of vibration, nerve velocity, proprioceptor feedback under skin receptor control, and can occur in static, dynamic and isokinetic muscle strength. This causes you to continue the preparations for the necessary evaluations in your postural stability and you watch. Particularly geriatrics reported that Otogo supports us to improve balance in us.

The purpose of this goal is to test in otago educational work on static and dynamic movements, lower hypertensive muscle work, capacity and capacity and competence.

DETAILED DESCRIPTION:
It is the ability to keep and maintain the body training balance control. Dynamic balance is the ability to maintain an individual's static position while the movement and posture are active while static. With aging, it is thought that the system will be applied in practice. Control of cerebral blood flow and synapse, which decreases with advanced age and hypertension, continues. In addition to slowing down in mental functions such as memory and learning, it progresses and accelerates in the sense of vibration, nerve velocity, proprioceptor feedback under skin receptor control, and can occur in static, dynamic and isokinetic muscle strength. This causes you to continue the preparations for the necessary evaluations in your postural stability and you watch.

Hypertension is defined as a systolic blood pressure of 140 mmHg and a diastolic blood pressure of 90 mmHg or more. The sudden decrease in blood flow as a result of sudden changes in blood pressure in Hypertension effects the mechanism in the control of postural balance.

Although there are studies to understand the relationship of hypertension with postural control and consequently the risk of falling, further studies are needed.

Current literature has reported that the balance program, which was developed to improve balance, especially in geriatric individuals, is effective. In this sense, the Otago Protocol: The Otago Exercise Program is an evidence-based, home-based, individually tailored strength and balance retraining program. The Otago Workout Program includes five strengthening exercises and 12 balance exercises. Participants are asked to do the exercises three times a week (starting with 10 repetitions). In addition, participants are asked to walk for 30 minutes 2 times a week (walking can be divided into days). Depending on the individual's strength and mobility, exercises can be advanced. It should be applied 3 times a week for an average of 1 hour.

The purpose of this goal is to test in Otago educational work on static and dynamic movements, lower hypertensive muscle work, capacity and capacity and competence.

Method Evaluation parameters Demographic Information Variables such as age, gender, height, weight, body mass index (BMI), dominant side, duration of education, medications used, pain, how long the symptoms are present if there is pain, exercise habits, and how long they sit during the day. will be saved.

Standardized Mini Mental Test It is a scale that can be applied easily and gives information about the degree of cognitive impairment. This test consists of subsections that assess orientation, registration, attention, calculation, recall, language tests, and configuration. The highest score that can be obtained from the test is 30 .

Muscle strength measurement of lower extremity The muscles of hip, knee and ankle circumference will be measured with a hand held digital dynamometer.

FAB-T balance survey This scale evaluates both the dynamic and static balance of the individual who will participate in the study with 10 questions in it, it is a balance test with a total of 40 points. If the participant achieves a score below 25 points, it indicates that the risk of falling is high. The Turkish reliability and validity study was conducted in May 2020 Posture Evaluation will be evaluated by the photography method.

Functional capacity:

To determine it, the participating individuals were asked to travel as far as they could walk for 6 minutes. Before the test, blood pressure, oxygen saturation, heart rate, walking distance, shortness of breath and fatigue level according to borg were evaluated. Immediately after the test, recovery (5 minutes later), the same values will be recorded again.

One-leg stand test (static balance) While the patient's eyes are open, hands on hips, feet are bare, and the hip is in a neutral position, care is taken to flex one knee and not to touch the flexed foot during the test. The time starts as soon as the foot is lifted from the ground and is recorded in seconds. 3 attempts are made for each foot and the best value is recorded.

Timed Sit and Stand Test:

The individual is asked to sit in a chair with back support with arms in front of the body and stand up. During the test, how long the individual sits and stands for 30 seconds is recorded. A score less than 10 indicates lower extremity weakness.

Timed Get Up and Walk Test: While the individual is sitting in a supported chair, he is asked to stand up and walk 3 meters and sit down again, and the time is recorded. A healthy individual is expected to complete it in 12 seconds.

International Survey of Physical Activity (IPAQ) It was developed to determine the physical activity levels of participants between the ages of 15-65. The validity and reliability study of IPAQ in Turkey (2005). Walking is the structure that separates the scores of moderate-intensity activities and vigorous activities. Walking requires knowing the duration (minutes) and frequency (days) of moderate activities and vigorous activities to calculate the total score. A score is obtained as "MET minute/week" by multiplying the minute, day and MET value. Physical activity levels; classified as low (<600 MET - min/week), moderate (600 - 3000 MET - min/week) and high (beneficial for health) (>3000 MET - min/week)(19)

Foot Function Index:

Foot function index; It consists of 23 items with 3 main subgroups as pain, disability and activity limitation. While the nine-item pain subscale measures the level of foot pain in various situations, the 9-item disability subscale determines the degree of difficulty in performing various functional activities due to foot problems. The activity limitation sub-scale, which includes five items, evaluates the activity limitations due to foot problems. Patients score all items with the Visual Analogue Scale (VAS) considering their foot conditions in the last 7 days.

Fall Activity Scale: It is a scale that asks the participants about 10 daily functions ranging from 1 to 10, 1 'I trust a lot' and 10 'I don't trust at all'. It was developed by Merry E. et al. in 1990. Turkish reliability and validity study was performed in 2009.

Training group: The Otago Protocol: The Otago Exercise Program is an evidence-based, home-based, individually tailored strength and balance retraining program. The Otago Workout Program includes five strengthening exercises and 12 balance exercises. Participants are asked to do the exercises three times a week (starting with 10 repetitions). In addition, participants are asked to walk for 30 minutes 2 times a week (walking can be divided into days). Depending on the individual's strength and mobility, exercises can be advanced. For example, adding hand weights to weight-lifting exercises or increasing repetitions. It should be applied 3 times a week for an average of 1 hour.

The training will last for 8 weeks and the evaluations will be evaluated before and after the training to determine the effectiveness of the training.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with HT (at least 6 months),
* Individuals who are independent in activities of daily living,

Exclusion Criteria:

* Those with neurological disease
* Those with Anxiety, Uncontrollable Hypertension, Chronic systemic disease

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
FAB-T balance survey | 10 minutes
  This scale evaluates both the dynamic and static balance of the individual who will participate in the study with 10 questions in it, it is a balance test with a total of 40 points. If the participant achieves a score below 25 points, it indicates that the risk of falling is high. The Turkish reliability and validity study was conducted by Iyigun et al. in May 2020 (15)

SECONDARY OUTCOMES:
Lower working muscle strength | 15 minutes
  The hip value and the muscles to be evaluated will be measured with a hand-held digital dynamometer.

OTHER OUTCOMES:
Functional capacity | 10 minutes
  In order to determine, the participating individuals were asked to attend the distance they can walk for 6 minutes. Pre-test blood pressure, oxygen saturation, heart rate, walking distance, dyspnea and fatigue level according to BORG were evaluated. Immediately after the test, recovery (after 5 min) the same values will be saved again
Stop Test on One Foot (Static Balance) | 10 minutes
  From the patient, the eyes are open hands in the hip, the feet are naked, while the flexion of flexion and flexion during the test during the test is cautioned to support the support. The time is started as soon as it is removed from the foot and is recorded. 3 trials are made for each foot and the best value is recorded
Time up and go test | 10 minutes
  The individual arms are asked to sit on a back-backed chair in front of the trunk. During the test, the individual is recorded to sit by 30 sec. Less than 10 score lower extremity is signal to strength

CONTACTS AND LOCATIONS:
Overall Officials: Necati Özler, Msc, Principal Investigator — nozler@eul.emu.tr
Locations (1):
- Necati Özler, Nicosia, Yeni Kent, Cyprus

IPD SHARING:
Plan to Share IPD: No